CLINICAL TRIAL: NCT05536271
Title: Pharmacogenetic Study of Bisoprolol in Egyptian Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BisoprololPG
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute coronary syndrome patients (Experimental): Acute coronary syndrome patients prescribed with bisoprolol
  Interventions: Drug: Bisoprolol Fumarate

INTERVENTIONS:
Drug: Bisoprolol Fumarate — antihypertensive medicine prescribed for acute coronary syndrome patients
  Other Names: concor

SUMMARY:
Acute coronary syndrome (ACS) is any group of clinical symptoms compatible with acute myocardial ischemia and includes unstable angina (UA), non-ST-segment elevation myocardial infarction (NSTEMI), and ST-segment elevation myocardial infarction (STEMI). (1). In Egypt, the overall prevalence of coronary heart disease (CHD) is 8.3 % (2). In addition, CHD in Egypt is the principal cause of death, responsible for 21.73% of total mortality (2).

Beta-blockers have shown to reduce the short-term risk of a reinfarction and the long-term risk of all-cause mortality and cardiovascular mortality (3). Beta blockers are used within 24 hours of ACS and given as long-term therapy after discharge (4). The Most frequently used drug in Egypt is bisoprolol.

In patients with myocardial infarction undergoing primary percutaneous coronary intervention, early intravenous betablocker before reperfusion reduced infarct size and increased left ventricular ejection fraction (4). Despite the established benefits of beta blockers in ACS (acute coronary syndrome patients), they showed interindividual variability in patient's' blood pressure and heart rate (5).

pharmacokinetic variability was found in bisoprolol response especially in elderly patients (6). Bisoprolol is eliminated in equal parts by hepatic metabolism by CYP2D6 and CYP3A4 enzymes and by the kidney(7). A possible cause for this variability may be due to CYP450 genetic polymorphism. The CYP450 activity ranges considerably within a population and includes ultrarapid metabolizers (UMs), extensive metabolizers (EMs), intermediate metabolizers (IMs) and poor metabolizers (PMs) (8).The proposed research in this application will investigate the correlation between CYP2D6 and CYP3A4 polymorphism and pharmacokinetics of bisoprolol and will investigate the impact of the Genes' polymorphism on the clinical effect of bisoprolol in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
1. Ethical committee approval will be obtained from Ethics committee of Faculty of Pharmacy, Damanhour University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. Over 100 patients diagnosed with acute coronary syndrome for whom bisoprolol therapy is prescribed , will be recruited from Alexandria university hospital.
4. whole blood samples will be collected for Analyses of CYP2D6 and CYP3A4 variant alleles.
5. Blood samples for plasma concentration measurements of bisoprolol will be drawn at steady-state peak levels after 2-4 hours of administration of bisoprolol.
6. Heart rate and blood pressure of the patients will be measured to assess the clinical effect of bisoprolol.
7. Echocardiogram will be obtained at baseline and after 1-3 months of therapy with bisoprolol to assess the effect of the drug on ventricular Remodeling.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted with chest pain suspected to have ACS (acute coronary syndrome).
2. Both with ST elevation (STEMI) and without ST elevation (N-STEMI ) and unstable angina.
3. HR > 50 bpm.
4. Systolic Blood pressure > 90 mmHg.

Exclusion Criteria:

Patients with contraindications to Bisoprolol therapy:

* Heart rate <60 bpm
* Systolic blood pressure <90 mmHg
* Moderate or severe left ventricular failure
* Shock
* heart block
* Active asthma/reactive airways disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
CYP2D6 gene polymorphism | 2 months
  CYP2D6 gene polymorphism
CYP3A5 gene polymorphism | 2 months
  CYP3A5 gene polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Sherouk Okda, Bachelor, Principal Investigator — Clinical Pharmacy Specialist, Damanhour University.; amira B kassem, PHD, Study Director — Lecturer of Clinical Pharmacy, Damanhour University.; ahmad salahaldin, PHD, Study Director — Lecturer of biochemisrty, Damanhour University.; ahmad alamrawy, PHD, Study Chair — cardiologist , alexandria university; noha ahmad, PHD, Study Chair — Lecturer of Clinical Pharmacy, Damanhour University.; sohila Alonsy, PHD, Study Chair — Lecturer of Analytical chemistry, Damanhour University.
Locations (1):
- Damanhour University, Damanhūr, Behira, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almahmeed W, Arnaout MS, Chettaoui R, Ibrahim M, Kurdi MI, Taher MA, Mancia G. Coronary artery disease in Africa and the Middle East. Ther Clin Risk Manag. 2012;8:65-72. doi: 10.2147/TCRM.S26414. Epub 2012 Feb 16. PMID 22368447
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Ibanez B, Macaya C, Sanchez-Brunete V, Pizarro G, Fernandez-Friera L, Mateos A, Fernandez-Ortiz A, Garcia-Ruiz JM, Garcia-Alvarez A, Iniguez A, Jimenez-Borreguero J, Lopez-Romero P, Fernandez-Jimenez R, Goicolea J, Ruiz-Mateos B, Bastante T, Arias M, Iglesias-Vazquez JA, Rodriguez MD, Escalera N, Acebal C, Cabrera JA, Valenciano J, Perez de Prado A, Fernandez-Campos MJ, Casado I, Garcia-Rubira JC, Garcia-Prieto J, Sanz-Rosa D, Cuellas C, Hernandez-Antolin R, Albarran A, Fernandez-Vazquez F, de la Torre-Hernandez JM, Pocock S, Sanz G, Fuster V. Effect of early metoprolol on infarct size in ST-segment-elevation myocardial infarction patients undergoing primary percutaneous coronary intervention: the Effect of Metoprolol in Cardioprotection During an Acute Myocardial Infarction (METOCARD-CNIC) trial. Circulation. 2013 Oct 1;128(14):1495-503. doi: 10.1161/CIRCULATIONAHA.113.003653. Epub 2013 Sep 3. PMID 24002794
- [Background] Agesen FN, Weeke PE, Tfelt-Hansen P, Tfelt-Hansen J; for ESCAPE-NET. Pharmacokinetic variability of beta-adrenergic blocking agents used in cardiology. Pharmacol Res Perspect. 2019 Jul 12;7(4):e00496. doi: 10.1002/prp2.496. eCollection 2019 Aug. PMID 31338197
- [Background] Taguchi M, Nozawa T, Igawa A, Inoue H, Takesono C, Tahara K, Hashimoto Y. Pharmacokinetic variability of routinely administered bisoprolol in middle-aged and elderly Japanese patients. Biol Pharm Bull. 2005 May;28(5):876-81. doi: 10.1248/bpb.28.876. PMID 15863897
- [Background] Tjandrawinata RR, Setiawati E, Yunaidi DA, Santoso ID, Setiawati A, Susanto LW. Bioequivalence study of two formulations of bisoprolol fumarate film-coated tablets in healthy subjects. Drug Des Devel Ther. 2012;6:311-6. doi: 10.2147/DDDT.S36567. Epub 2012 Oct 30. PMID 23139624
- [Background] Mohammed Alkreathy H, Mohammed Eid Alsayyid K, Alaama JY, Al Ghalayini K, Karim S, Esmat A, Damanhouri ZA. Bisoprolol responses (PK/PD) in hypertensive patients: A cytochrome P450 (CYP) 2D6 targeted polymorphism study. Saudi J Biol Sci. 2020 Oct;27(10):2727-2732. doi: 10.1016/j.sjbs.2020.06.022. Epub 2020 Jun 20. PMID 32994732